CLINICAL TRIAL: NCT02233218
Title: A Phase 1, Open Label, Non-randomized, Two-cohort, Single-sequence, Crossover Study to Investigate the Pharmacokinetic Drug-drug Interaction and Safety of Telmisartan/Amlodipine and Rosuvastatin in Healthy Male Volunteers
Brief Title: The Pharmacokinetic Drug-drug Interaction and Safety of Telmisartan/Amlodipine and Rosuvastatin in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: YH22189-101
Record Dates: First submitted 2014-08-26; First posted 2014-09-08 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Healthy Male Volunteer
MeSH Terms: interventions — Telmisartan; Amlodipine; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- telmisartan, Amlodipine, Rosuvastatin (Experimental): This arm is consist of 40 subjects. Telmisartan80mg + Amlodipine 10mg 9 days, Telmisartan80mg + Amlodipine 10mg , Rosuvastatin 20mg 5days Total 14days administration of investigational products to healthy male volunteers
  Interventions: Drug: Telmisartan; Drug: Amlodipine; Drug: Rosuvastatin
- Telmisartan, Amlodipine, Rosuvastatin (Experimental): This arm is consist of 20 subjects. Rosuvastatin 20mg 5 days, Rosuvastatin 20mg , Telmisartan80mg + Amlodipine 10mg 9days, Total 14days administration of investigational products to healthy male volunteers
  Interventions: Drug: Telmisartan; Drug: Amlodipine; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Telmisartan
Drug: Amlodipine
Drug: Rosuvastatin

SUMMARY:
To investigate the pharmacokinetic Drug-drug interaction

DETAILED DESCRIPTION:
The purpose of this study is to investigate the pharmacokinetic Drug-Drug(telmisartan, amlodipine and/ or rosuvastatin) interaction and safety in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers aged 19 to 50
2. Participant who has a body weight that is >=55kg(male) and body mass index (BMI) level that is 18~30
3. Provision of signed written informed consent

Exclusion Criteria:

1. History of clinically significant disease
2. History of clinically significant hypersensitivity or hypersensitivity reactions to drugs and other medications (aspirin, antibiotics, etc.), including components such as Telmisartan, Rosuvastatin and Amlodipine
3. A history of drug abuse or the presence of positive reactions to drugs that have abuse potential in urine screenings for drugs
4. Administration of other investigational products within 2 months prior to the first dosing.
5. Administration of herbal medicine within 2 weeks or administration of ethical drugs within 2 weeks or administration of over-the-counter (OTC) drugs within 1 week prior to the first dosing of the investigational product (if the investigator (study doctor) determines that the person meets other criteria appropriately, the relevant person may participate in the study)
6. Volunteers considered not eligible for the clinical trial by the investigator (study doctor) due to the reasons including laboratory test results, ECGs, or vital signs.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Area under the plasma/serum/blood drug concentration-time curve in steady-state of Telmisartan and Amlodipine | 0h~24hr at Day 9 (when is expected the steady state of Telmisartan and Amlodipine) and 0~24hr at Day 14 (when is expected the steady state of Telmisartan, Amlodipine and Rosuvastatin)
Maximum concentration of drug in plasma/serum/blood in steady-state of Telmisartan and Amlodipine | 0h~24hr at Day 9 (when is expected the steady state of Telmisartan and Amlodipine) and 0~24hr at Day 14 (when is expected the steady state of Telmisartan, Amlodipine and Rosuvastatin)
Area under the plasma/serum/blood drug concentration-time curve in steady-state of Rosuvastatin | 0h~24hr at Day 5 (when is expected the steady state of Rosuvastatin) and 0~24hr at Day 14 (when is expected the steady state of Telmisartan, Amlodipine and Rosuvastatin)
Maximum concentration of drug in plasma/serum/blood in steady-state of Rosuvastatin | 0h~24hr at Day 5 (when is expected the steady state of Rosuvastatin) and 0~24hr at Day 14 (when is expected the steady state of Telmisartan, Amlodipine and Rosuvastatin)

SECONDARY OUTCOMES:
Time of peak concentration in steady state of Telmisartan and Amlodipine | 0h~24hr at Day 9 (when is expected the steady state of Telmisartan and Amlodipine) and 0~24hr at Day 14 (when is expected the steady state of Telmisartan, Amlodipine and Rosuvastatin)
Minimum concentration of drug in plasma/serum/blood in steady-state of Telmisartan and Amlodipine | 0h~24hr at Day 9 (when is expected the steady state of Telmisartan and Amlodipine) and 0~24hr at Day 14 (when is expected the steady state of Telmisartan, Amlodipine and Rosuvastatin)
Area under the plasma/serum/blood drug concentration-time curve in steady-state of N- desmethyl rosuvastatin | 0h~24hr at Day 5 (when is expected the steady state of Rosuvastatin) and 0~24hr at Day 14 (when is expected the steady state of Telmisartan, Amlodipine and Rosuvastatin)
Maximum concentration of drug in plasma/serum/blood in steady-state of N- desmethyl rosuvastatin | 0h~24hr at Day 5 (when is expected the steady state of Rosuvastatin) and 0~24hr at Day 14 (when is expected the steady state of Telmisartan, Amlodipine and Rosuvastatin)
Time of peak concentration in steady state of rosuvastatin and N- desmethyl rosuvastatin | 0h~24hr at Day 5 (when is expected the steady state of Rosuvastatin) and 0~24hr at Day 14 (when is expected the steady state of Telmisartan, Amlodipine and Rosuvastatin)
Minimum concentration of drug in plasma/serum/blood in steady-state of Rosuvastatin and N- desmethyl rosuvastatin | 0h~24hr at Day 5 (when is expected the steady state of Rosuvastatin) and 0~24hr at Day 14 (when is expected the steady state of Telmisartan, Amlodipine and Rosuvastatin)

CONTACTS AND LOCATIONS:
Overall Officials: Minkgyu Park, Ph.D, M.D., Principal Investigator — Dong-A university hospital of Korea
Locations (1):
- Dong-A university hospital, Pusan, South Korea